CLINICAL TRIAL: NCT01650194
Title: A Phase 2 Study Determining Safety and Tolerability of Enzalutamide (Formerly MDV3100) in Combination With Abiraterone Acetate in Bone Metastatic Castration-Resistant Prostate Cancer Patients
Brief Title: A Study to Determine Safety and Tolerability of Enzalutamide (MDV3100) in Combination With Abiraterone Acetate in Bone Metastatic Castration-Resistant Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0011
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: abiraterone acetate; prednisone; enzalutamide; cancer; prostate; MDV3100
MeSH Terms: conditions — Neoplasms | interventions — enzalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide + Abiraterone + Prednisone (Experimental): Participants received enzalutamide combined with abiraterone acetate once daily plus prednisone twice daily.
  Interventions: Drug: enzalutamide; Drug: abiraterone acetate; Drug: prednisone

INTERVENTIONS:
Drug: enzalutamide — Participants received 160 mg of enzalutamide orally once daily (4 capsules, 40 mg each).
  Other Names: MDV3100
Drug: abiraterone acetate — Participants received 1000 mg of abiraterone acetate orally once daily (4 tablets, 250 mg each).
Drug: prednisone — Participants received 5 mg of prednisone orally twice daily (2 tablets, 5 mg each).

SUMMARY:
The purpose of this study was to explore the safety and tolerability of enzalutamide in combination with abiraterone acetate plus prednisone. Subjects diagnosed with cancer of the prostate that was getting worse and spreading to the bone despite receiving hormone treatment were enrolled and received study treatment until disease progression.

DETAILED DESCRIPTION:
For the study duration, all subjects maintained androgen deprivation with a gonadotropin releasing hormone (GnRH) agonist or antagonist or orchiectomy. Study drug was administered until disease progression. Disease progression was defined as a composite endpoint consisting of either clinical deterioration, radiographic progression or prostate-specific antigen (PSA) progression according to the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Presence of metastatic disease to the bone
* Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration)
* Subject receiving bisphosphonate or denosumab therapy must have been on stable doses for at least 4 weeks prior to Day 1
* Progressive disease defined as one or more of the following three criteria (Note: subjects who received an antiandrogen must demonstrate disease progression following discontinuation of antiandrogen):

  * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the Screening visit should be ≥ 2 ng/mL
  * Soft tissue disease progression as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
  * Bone disease progression defined by PCWG2 criteria (two or more new lesions on bone scan compared with prior scan)
* Subject previously treated with chemotherapy must have no more than two prior chemotherapy regimens for the treatment of metastatic prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Agree to use a double-barrier method of contraception which involves the use of a condom in combination with one of the following: contraceptive sponge, diaphragm, or cervical ring with spermicidal gel or foam, if having sex with a woman of child-bearing potential during the length of the study and for one week after abiraterone is discontinued and for at least three months after enzalutamide is discontinued
* Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Known or suspected metastases in the brain
* Absolute neutrophil count < 1,000/μL, platelet count < 75,000/μL, and hemoglobin < 9 g/dL (NOTE: subject may not have received any growth factors or blood transfusions within seven days of the hematologic laboratory values obtained at the Screening visit)
* Total bilirubin (TBL), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal
* Creatinine (Cr) > 2 mg/dL
* Treatment with androgen receptor antagonists (bicalutamide, flutamide, nilutamide), 5-α reductase inhibitors (finasteride, dutasteride), estrogens, chemotherapy, or biologic therapy within 4 weeks of Day 1 visit
* Radiation therapy within 3 weeks (if single fraction of radiotherapy within 2 weeks) of Day 1 visit, or radionuclide therapy within 8 weeks of Day 1
* Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
* Structurally unstable bone lesions suggesting impending fracture
* History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases, or alcoholism. Also, history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Day 1 visit)
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months of Screening visit;
  * Uncontrolled angina within 3 months of Screening visit;
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months of the Screening visit results in a left ventricular ejection fraction that is ≥ 45%
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes)
  * Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on the Electrocardiogram (ECG) > 470 msec.
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  * Hypotension (systolic blood pressure < 86 mmHg or bradycardia with a heart rate of <50 beats per minute on the ECG., unless pharmaceutically induced and thus reversible (i.e. beta blockers).
  * Uncontrolled hypertension as indicated by a resting systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg
* Prior use of ketoconazole, abiraterone acetate or enzalutamide, or participation in a previous clinical trial of ketoconazole, abiraterone acetate or enzalutamide
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) of Screening visit
  * History of GI bleeding within 6 months of Screening visit
* Active or symptomatic viral hepatitis or chronic liver disease
* Known history of pituitary or adrenal dysfunction

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Site US2492 MD Anderson Cancer Ctr, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Assi R, Temraz S, Shamseddine A, Mukherji D. New Compounds Targeting the Androgen Receptor for Treatment of Advanced Prostate Cancer. Curr Drug Targets. 2016;17(3):290-302. doi: 10.2174/1389450116666150907101044. PMID 26343110
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants in this all male study were enrolled at 1 site in the United States (US).
Pre-assignment Details: All eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled. A total of 64 participants were screened for eligibility.
Period: Overall Study
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Started | 60
Treated | 60
Completed | 13
Not Completed | 47
Not completed — Progressive Disease (PD) | 35
Not completed — Withdrawal by Subject | 2
Not completed — Miscellaneous | 10

BASELINE CHARACTERISTICS:
Population: The analysis population for all baseline measures consisted of all participants who were enrolled in the study.
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51
  Black or African American | 6
  Asian | 2
  Other | 1
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 57
  Hispanic or Latino | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event occurring or worsening between the start of study treatment date and the latest date of 30 days after the last dose date or the 30-day follow-up visit date, and not later than the data cut-off date or the date of death. AEs, including abnormal clinical laboratory values, were graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) guidelines (V4.03).
Time Frame: From the first dose of study drug administration up 30 days following the last dose of study drug date, with a median duration of treatment of 10.1 months.
Population: The analysis population consisted of the safety analysis set (SAF) which consisted of all participants who received at least 1 dose of any drug of the study combination treatment (i.e., enzalutamide, abiraterone and prednisone).
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 60
Participants
  Any TEAE | 60
  Enzalutamide-related TEAEs | 56
  Abiraterone-related TEAEs | 58
  Prednisone-related TEAEs | 16
  Deaths | 0
  Serious TEAEs | 10
  Enzalutamide-related serious TEAEs | 0
  Abiraterone-related serious TEAEs | 2
  Prednisone-related serious TEAEs | 0
  TEAEs leading to discontinuation of enzalutamide | 3
  Enza-related TEAEs leading to disc. of enza | 0
  Abiraterone-related TEAEs leading to disc. of enza | 0
  Prednisone-related TEAEs leading to disc. of enza | 0
  TEAEs leading to discontinuation of abiraterone | 1
  Abiraterone-related TEAEs leading to disc. of abi | 1

2. Secondary Outcome: Change From Baseline in Testosterone Concentration in Bone Marrow Aspirate
Description: Testosterone concentration in bone marrow aspirate was measured by laboratory results derived from bone marrow samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the biomarker testosterone evaluable set (BTES) which consisted of all participants from the SAF with baseline and week 9 testosterone laboratory results derived from bone marrow samples.
Measure: Geometric Mean (Standard Deviation); unit: pmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 45
pmol/L | -19.48 (257.923)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Testosterone biomarker results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p = 0.6150, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Dihydrotestosterone (DHT) Concentration in Bone Marrow Aspirate
Description: DHT concentration in bone marrow aspirate was to be measured by laboratory results derived from bone marrow samples processed through liquid chromatography mass spectrometry. DHT bone data were not collected.
Time Frame: Baseline and Week 9
Population: DHT bone data were not collected.
Groups:
- Enzalutamide + Abiraterone + Prednisone: Participants received enzalutamide combined with abiraterone acetate once daily plus prednisone twice daily. DHT bone data were not collected.
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Cortisol in Bone Marrow Aspirate
Description: Cortisol in bone marrow aspirate was measured by laboratory results derived from bone marrow samples.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the biomarker cortisol evaluable set (BCES) which consisted of all participants from the SAF with baseline and week 9 cortisol laboratory results derived from bone marrow samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 47
nmol/L | -46.86 (48.022)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Cortisol biomarker results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Androstenedione in Bone Marrow Aspirate
Description: Androstenedione in bone marrow aspirate was measured by laboratory results derived from bone marrow samples.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the biomarker androstenedione evaluable set (BAOS) which consisted of all participants from the SAF with baseline and week 9 androstenedione laboratory results derived from bone marrow samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 37
nmol/L | -0.32 (0.342)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Androstenedione biomarker results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Progesterone in Bone Marrow Aspirate
Description: Progesterone in bone marrow aspirate was measured by laboratory results derived from bone marrow samples.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the biomarker progesterone evaluable set (BOES) which consisted of all participants from the SAF with baseline and week 9 progesterone laboratory results derived from bone marrow samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 41
nmol/L | 1.16 (1.104)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Progesterone biomarker results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Pregnenolone in Bone Marrow Aspirate
Description: Pregnenolone in bone marrow aspirate was measured by laboratory results derived from bone marrow samples.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the biomarker pregnenolone evaluable set (BEES) which consisted of all participants from the SAF with baseline and week 9 pregnenolone laboratory results derived from bone marrow samples.
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 42
pg/ml | 1381.44 (1513.324)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Pregnenolone biomarker results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Testosterone Concentration in Blood
Description: Testosterone concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the plasma testosterone evaluable set (PTES) which consisted of all participants from the SAF with baseline and week 9 testosterone laboratory results derived from plasma samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 49
nmol/L | -0.06 (0.068)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Testosterone blood results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in DHT Concentration in Blood
Description: DHT concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry. The endpoint could not be analyzed since no participants had DHT levels over the lower limit of quantification (LLOQ).
Time Frame: Baseline and Week 9
Population: The endpoint could not be analyzed since no participants had DHT levels over the LLOQ.
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Cortisol Concentration in Blood
Description: Cortisol concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the plasma cortisol evaluable set (PCES) which consisted of all participants from the SAF with baseline and week 9 cortisol laboratory results derived from plasma samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 52
nmol/L | -48.81 (43.725)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Cortisol blood results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Androstenedione Concentration in Blood
Description: Androstenedione concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the plasma androstenedione evaluable set (PAOS) which consisted of all participants from the SAF with baseline and week 9 androstenedione laboratory results derived from plasma samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 37
nmol/L | -0.24 (0.206)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Androstenedione blood results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Progesterone Concentration in Blood
Description: Progesterone concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the plasma progesterone evaluable set (POES) which consisted of all participants from the SAF with baseline and week 9 progesterone laboratory results derived from plasma samples.
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 48
nmol/L | 1.43 (2.434)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Progesterone blood results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p = 0.0002, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Pregnenolone Concentration in Blood
Description: Pregnenolone concentration in blood was measured by laboratory results derived from plasma samples. Plasma samples were derived from collected blood samples processed through liquid chromatography mass spectrometry.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the plasma pregnenolone evaluable set (PEES) which consisted of all participants from the SAF with baseline and week 9 pregnenolone laboratory results derived from plasma samples.
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 47
pg/ml | 1507.42 (1699.335)
Statistical Analysis 1: Comparison: Enzalutamide + Abiraterone + Prednisone; Pregnenolone blood results collected at baseline and at Week 9 were compared using the paired t-test to evaluate the effect of enzalutamide; Test type: Other; p < .0001, t-test, 2 sided

14. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Prostate-Specific Antigen (PSA) Levels
Description: Prostate-specific antigen progression by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) was defined as a PSA increase ≥25% and ≥2 ng/ml above the post-baseline nadir, and which was confirmed by the first subsequent value of 3 or more weeks later.
Time Frame: Baseline and EoT; the median duration of treatment was 10.1 months.
Population: The analysis population consisted of the SAF (participants with available data).
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 59
ug/L | 36.35 (444.355)

15. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured as the time from the date of first dose of any drug of the study combination treatment until the first evidence of documented progression (a composite endpoint consisting of radiographic progression or PSA progression by PCWG2 or clinical deterioration) or death in the absence of progression (whichever came first) or the date last known to be progression free. The Kaplan-Meier (KM) 95% CI was based on Brookmeyer and Crowley robust non-parametric method.
Time Frame: Up to 1849 days
Population: The analysis population consisted of the SAF.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 60
days | 251 [147.0 to 337.0]

16. Secondary Outcome: Percentage of Participants With Objective Response for Soft Tissue Lesions According to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST)
Description: Objective response was based on RECIST version 1.1 for soft tissue lesion on Magnetic resonance imaging (MRI) / Computerized tomography (CT) and the PCWG2 guidelines for bone lesions on bone scans and was defined as partial response (PR) or complete response (CR) based on the investigators' assessments of target, non-target and new lesions while on study treatment. The 95% for objective response rate was based on exact binomial 95% confidence interval (Clopper-Pearson).
Time Frame: Up to 1849 days
Population: The analysis population consisted of the SAF (participants with measurable soft tissue disease per RECIST 1.1 at baseline with available data).
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 16
percentage of participants | 68.8 [41.3 to 89.0]

17. Secondary Outcome: Bone Scan Response at EoT
Description: PD: ≥1 of 3 criteria: PSA progression: ≥2 rising PSA levels, interval of ≥1 week between each determination. Soft tissue disease progression: RECIST 1.1. Bone disease progression: PCWG2 criteria (≥2 or new lesions on bone scan compared with prior scan). Target lesion CR: disappearance of all target lesions, PR as ≥30% decrease in sum of longest diameter (LD) of target lesions, referencing baseline sum LD, SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, referencing smallest sum LD since treatment start, PD ≥20% increase in sum of LD of target lesions, referencing smallest sum LD recorded since treatment start or appearance of ≥1 new lesions. Non-target lesions CR: disappearance of all non-target lesions and normalization of tumor marker level, SD: persistence of ≥1 non-target lesions and/or maintenance of tumor marker level above normal limits, PD: appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: EoT; the median duration of treatment was 10.1 months.
Population: The analysis population consisted of the SAF (participants with available data).
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 52
Participants
  Complete Response (CR) | 1
  Progressive Disease (PD) | 15
  Non-CR/Non-PD | 35
  Not Evaluable | 1

18. Secondary Outcome: Change From Baseline to EoT in Bone Specific Alkaline Phosphatase
Description: Bone metabolism marker bone specific alkaline phosphatase levels were derived from blood samples collected.
Time Frame: Baseline and EoT; the median duration of treatment was 10.1 months.
Population: The analysis population consisted of the SAF (participants with available data).
Measure: Geometric Mean (Standard Deviation); unit: ug/L
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 49
ug/L | -5.18 (43.626)

19. Secondary Outcome: Change From Baseline in Urine N-Telopeptide
Description: Bone metabolism marker urine N-telopeptide levels were derived from urine samples collected.
Time Frame: Baseline and Week 9
Population: The analysis population consisted of the SAF (participants with available data).
Measure: Geometric Mean (Standard Deviation); unit: nmolBCE/mmolcreat
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 34
nmolBCE/mmolcreat | 29.35 (85.927)

20. Other Pre Specified Outcome: Androgen Receptor Signaling Assessed by Expression and Localization of Androgen Receptor (AR), CYP17 Expression, Splice Variants, and Pathways Linked With Non-classical AR Signaling and Bone Development
Description: The endpoint was considered exploratory and no analysis was planned.
Time Frame: Baseline and Week 9
Population: Data for these endpoints were not collected.
Arm/Group | Enzalutamide + Abiraterone + Prednisone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up 30 days following the last dose of study drug date, with a median duration of treatment of 10.1 months.
Arm/Group | Enzalutamide + Abiraterone + Prednisone
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 9/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Abiraterone + Prednisone (N=60)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Macular oedema (Eye disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Abiraterone + Prednisone (N=60)
Anaemia (Blood and lymphatic system disorders) | 21 (40)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 9 (14)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 14 (28)
Vomiting (Gastrointestinal disorders) | 6 (20)
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 43 (62)
Influenza like illness (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 9 (13)
Pyrexia (General disorders) | 7 (8)
Herpes zoster (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 9 (12)
Joint injury (Injury, poisoning and procedural complications) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 8 (10)
Alanine aminotransferase increased (Investigations) | 18 (70)
Aspartate aminotransferase increased (Investigations) | 22 (54)
Blood albumin decreased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 32 (64)
Blood bilirubin increased (Investigations) | 12 (26)
Blood creatinine increased (Investigations) | 3 (5)
Blood glucose increased (Investigations) | 5 (7)
Blood magnesium decreased (Investigations) | 6 (8)
Blood potassium decreased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 6 (12)
Neutrophil count decreased (Investigations) | 7 (8)
Platelet count decreased (Investigations) | 7 (12)
White blood cell count decreased (Investigations) | 14 (22)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 41 (96)
Hypernatraemia (Metabolism and nutrition disorders) | 7 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (20)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (28)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (19)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (18)
Balance disorder (Nervous system disorders) | 3 (4)
Cognitive disorder (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 8 (9)
Headache (Nervous system disorders) | 11 (17)
Memory impairment (Nervous system disorders) | 6 (7)
Paraesthesia (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 3 (5)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (7)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flush (Vascular disorders) | 27 (39)
Hypertension (Vascular disorders) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2014-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT01650194/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT01650194/SAP_001.pdf